CLINICAL TRIAL: NCT00806975
Title: Randomized，Open-Label，2-Period，Crossover Comparison of Randomized，Open-Label，2-Period，Crossover Comparison of Novo Rapid 30 Mix Injection FlexPen® and Humalog 25 Mix Injection KwikPen® in Adult Patients With Type 2 Diabetes Mellitus
Brief Title: Comparison of Novo Rapid 30 Mix Injection FlexPen® and Humalog 25 Mix Injection KwikPen® in Type 2 Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nagaoka Red Cross Hospital (Other)
Responsible Party: Kyuzi Kamoi, Nagaoka Red Cross Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2008-12-09; First posted 2008-12-11 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Diabetes Complications; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- usability and preference (Other)
  Interventions: Device: KwikPen® and FlexPen®

INTERVENTIONS:
Device: KwikPen® and FlexPen® — The treatment is changed to twice a day injection of the same unit of Novo Rapid 30 Mix injection FlexPen® or Humalog Mix 25 injection KwikPen®for 3 months, after which the final assessment is made.

SUMMARY:
The purpose of this study is to investigate patient's usability, preference and blood glucose control for the new prefilled disposable insulin lispro mixture (Humalog Mix 25 injection KwikPen®). For that purpose, randomized open-label, 2-period direct comparative crossover study is planned in comparison with insulin aspart mixture (Novo Rapid 30 Mix injection FlexPen®).

DETAILED DESCRIPTION:
* Concomitant drugs The treatment with other insulin preparation is prohibited during the study period. As to the drugs except insulin that have been used for the treatment of diabetes and its complication since the time before the study, the content should not be changed during the study in principle unless the complication is cured. If any new complication occurs during the study period, an appropriate treatment is given by the judgment of investigator.
* Compliance with treatment method The investigator gives sufficient explanation on the following contents to the patient.

  * To inject the prescribed volume of insulin at the prescribed time.
  * To observe the appointed date for the next visit.
* Termination of assessment The study is discontinued if any of the following events occurs after the start of study.

  * Important protocol violation
  * When continued treatment is judged difficult due to the onset of an adverse event
  * Death
  * When the follow-up of patient becomes impossible
  * Other than the above, when the investigator judges it necessary to discontinue the study

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus patients
* Patients who have used Humalog Mix 25 injection KwikPen® or Novo Rapid 30 Mix injection FlexPen® for 3 months or more.
* Outpatients regularly visiting hospital
* Patients 20 years old or older but under 80 years old (gender is disregarded)

Exclusion Criteria:

* Patients with a serious complication in the heart, liver or kidney
* Pregnant or possibly pregnant patients, or lactating patients
* Patients complicated with a malignant tumor at present.
* Patients allergic to insulin analog preparations.
* Patients taking an illegal drug.
* Patients participating in other clinical study.
* Other than the above, patients judged inappropriate as the subjects of this study by the investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
HbA1c change rate from the start to 12 and 24 weeks are investigated and compared. Furthermore, using a questionnaire sheet "IDSQ-J" related to the insulin infusion device, the patient's usability and satisfaction with KwikPen® or FlexPen® are performed. | 24 weeks

SECONDARY OUTCOMES:
As the secondary endpoints, the incidence of hypoglycemia, changes in body weight (BMI) and blood pressure, and the dose of insulin are investigated and compared before and after the changeover. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyuzi Kamoi, MD, Study Director — Nagaoka Red Cross Hospital
Locations (1):
- Nagaoka Red Cross Hospital, 2-291 Nagaoka, Niigata, Japan